CLINICAL TRIAL: NCT00426634
Title: Head-Off Environmental Asthma in Louisiana
Brief Title: Children With Asthma in New Orleans After Hurricane Katrina
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Collaborators: Merck Childhood Asthma Network (MCAN) (Unknown)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999907068; 07-E-N068
Record Dates: First submitted 2007-01-24; First posted 2007-01-25 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2016-08-30

CONDITIONS: Asthma; Allergies
Keywords: Asthma; Allergens; Mold; Asthma Counselor; Environmental Remediation
MeSH Terms: conditions — Asthma; Hypersensitivity

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will examine whether exposure to the increased levels of mold and other allergens in New Orleans post-Hurricane Katrina affect symptoms in children with asthma. It will also determine if having an asthma counselor (AC) can reduce a child s asthma symptoms in this setting. An AC helps the families in the study obtain appropriate health care, medicines and social services for their asthmatic child and instructs them about avoiding allergens and ridding allergens from the home.

Children between 4 and 12 years of age living in Orleans Parish or surrounding areas impacted by flooding who have moderate to severe asthma may be eligible for this study.

Parents provide a family medical history and information about the child s asthma symptoms, medications and medical history. The children undergo the following procedures:

* Medical examination and blood tests
* Spirometry (for children 6 and older) or peak flow (for children under 6) test: For spirometry, the child wears a nose clip and breathes into a mouthpiece attached to a machine that measures how fast air moves out of the child s lungs. For the peak flow meter test, the child blows into a plastic tube after taking a deep breath.
* Allergy skin testing: 24 common allergens are applied to the arm by little pricks or scratches and the skin is observed for reactions to the allergens.

Study staff visit the participants homes three times during the 1-year study to test for moisture, mold and other allergens. After the first visit, families are randomly assigned to one of two groups. Group 1 participants attend two educational group sessions about asthma and then three individual sessions. An AC visits the home one time during the study to instruct the family on how to use supplies provided to reduce allergens in the home. Group 2 participants have an individual special teaching meeting with the AC at the end of the study. After the meeting, the AC visits the home to instruct the family on use of the supplies.

Families are surveyed by phone every 3 months during the study to answer questions about the child s asthma attacks, medicines used, doctor visits, school days, missed, or work days missed to care for the child. At the end of the study, the child has a final medical examination, blood test, and breathing test.

DETAILED DESCRIPTION:
This document presents the protocol for conducting the Head-off Environmental Asthma in Louisiana (HEAL) study in New Orleans, Louisiana. The goal of the HEAL study is to implement and test an Asthma Counselor (AC) intervention program that addresses the multidimensional impact of hurricane Katrina on children with asthma in New Orleans. HEAL is a prospective, controlled trial in which children will be randomly assigned to one of two treatment groups. Group 1 children will receive an AC intervention focused on case management, adherence to medications and education on allergen avoidance. The responsibilities of the AC in this study are enhanced relative to previous initiatives such as the National Cooperative Inner City Asthma Study (NCICAS) AC intervention to also provide families with education aimed at reducing mold, allergens, and moisture in their homes, and materials to aid this effort (dehumidifiers and HEPA air filters). Since 90% of children with asthma in New Orleans are sensitive to dust allergens, established allergen control measures will be incorporated into the AC intervention as well. Group 2 children will receive a high quality standard of care based on the National Asthma Education and Prevention Program (NAEPP)-NIH guidelines. An abbreviated AC intervention will be provided to children in Group 2 at the conclusion of the study. Both treatments will be administered over a 12-month period during which the children in both groups will receive an extensive clinical evaluation (at baseline and 12-months) and three environmental home evaluations (focused on moisture, mold and other allergens). In addition to monitoring the effectiveness of the AC at environmental remediation education, the environmental home evaluations will also allow some characterization of the relationships between allergens, post-Katrina environmental exposures and asthma morbidity.

In addition to the enhanced AC intervention, a separate school based survey will be administered to a sample population of children to examine asthma prevalence and assess living conditions and stress levels that may have been influenced by hurricane Katrina. The survey population will consist of a sample of the families of Orleans Parish school children stratified by age, schools and geographic area of the Parish. The results of the survey, in combination with the results of the AC intervention, will give us an overview of the extent and severity of the asthma problem in post hurricane Katrina New Orleans.

The HEAL project is a collaborative multi-institutional research project conducted by the Tulane University School of Public Health and Tropical Medicine and the New Orleans Department of Health. To support those efforts, Rho, Inc. will provide for coordination of data and study activities.

ELIGIBILITY:
* INCLUSION CRITERIA:

A child will be included in the HEAL intervention study if he or she:

1. Is a male or female child four to twelve years old, inclusive, at the time of recruitment, living in Orleans Parish or surrounding areas impacted by flooding.
2. Has previously been given a diagnosis of asthma by a healthcare provider and who has symptoms as described below (Criteria 3) for more than one year.
3. Is currently receiving long-term asthma control therapy, as reported at baseline, and either has symptoms consistent with persistent asthma (criterion 3a, see below) or has evidence of uncontrolled disease (criterion 3b); or is not currently receiving long-term asthma control therapy and has symptoms consistent with persistent asthma (criterion 3a) and also has evidence of uncontrolled disease (criterion 3b):

3a. Evidence of persistent asthma as defined by the National Asthma Education and Prevention Program (NAEPP) of the National Heart Lung and Blood Institute Expert Panel Report 2: Guidelines for the Diagnosis and Management of Asthma (1997), which includes: asthma symptoms 3 or more days per week during the last two weeks, sleep disturbed due to asthma at least 3 times in the past month, or albuterol use (Metered Dose Inhaler or nebulizer) for quick relief at least 8 times in the past two weeks, not including use as a preventive for exercise.

3b. Evidence of uncontrolled disease as defined by at least one of the following additional criteria:

i. One asthma-related unscheduled visit to an emergency department (ED), urgent care (UC), or clinic in the previous 12 months.

ii. One asthma-related overnight hospitalization in the previous 12 months.

iii. One or more bursts of oral corticosteroids or equivalent in the previous 12 months.

4) Has a parent or legal guardian willing to sign the written informed consent prior to initiation into the study.

5) Is willing to sign the assent form, if age appropriate.

EXCLUSION CRITERIA:

A child will be excluded from the HEAL intervention study if she or he:

1. Is defined as having mild intermittent asthma at baseline evaluation.
2. Has had a life-threatening asthma exacerbation in the last 5 years requiring intubation, mechanical ventilation, or resulting in a hypoxic seizure.
3. Has significant medical illnesses other than asthma such as: any hematologic, endocrine, respiratory (other than asthma) or cardiac condition requiring daily medications; significant neurological disorder requiring daily medications; any clotting disorder; any obvious severe mental retardation that prohibits the child or the child s caregiver from answering questions or following instructions; any autoimmune disease; any immune deficiency; or any other serious medical condition including Juvenile diabetes mellitus, hypo- or hyper- thyroidism, hemophilia, Von Willebrands disease, sickle cell disease, cerebral palsy, rheumatoid arthritis, lupus, psoriasis, hyperimmunoglobulin E syndrome, or diagnosed allergic bronchopulmonary aspergillosis.
4. Has not had a home evaluation completed within 4-6 weeks of the Screening Visit (may be re-screened).
5. Lives with a foster parent.
6. Has caregiver (typically the parent or guardian) who does not have access to a phone.
7. Plans to move out of the recruitment area over the next year.

One child from each household will be selected to participate in the study. In the case of multiple eligible children, the youngest child will be included in the study.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2007-01-19; Study Completion 2016-08-30

CONTACTS AND LOCATIONS:
Overall Officials: Triesta M Fowler-Lee, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- Tulane University Health Sciences Center, New Orleans, Louisiana, United States